CLINICAL TRIAL: NCT06523348
Title: Ultrasound of the Quadriceps Femoris for the Diagnosis of Frailty in the Intensive Care Unit, Compared With the Clinical Frailty Scale (CFS)
Brief Title: Ultrasound of the Quadriceps Femoris Compared With the Clinical Frailty Scale
Acronym: QUADRI-REA
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0180; N° ID-RCB (Other: 2024-A01052-45)
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Frailty; Intensive Care Unit Syndrome
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: quadricipital muscle ultrasound — ultrasound depth measurement of the quadriceps muscle

SUMMARY:
This is a single-centre prospective diagnostic study. When a patient is admitted to the inclusion centre, the clinician responsible for the patient checks the inclusion and exclusion criteria. The no objection from the patient (or their trusted support person or, failing that, a close if the patient is unable to give consent) is sought.The CFS scale is completed and recorded by the clinician in the observation observation notebook.The clinician performs a quadricipital muscle ultrasound, specifically for research purposes, with no changes to the therapeutic and its results are recorded in the observation notebook.

observation notebook.At 3 months after inclusion, information was collected from the medical records to identify secondary endpoints.

Translated with DeepL.com (free version)

DETAILED DESCRIPTION:
Fragility is defined as a decline in physical and mental capacities leading to increased vulnerability to pathologies. It is now accepted that frail patients have a higher morbidity and mortality rate than non-frail patients. In intensive care, the prevalence of frail patients reaches 30% of patients admitted. These patients have a higher rate of complications and mortality than non-fragile patients.Identifying frail patients is therefore a major challenge in the ICU, to enable the risk of short-term mortality to be stratification of the risk of mortality in the short, medium and long term, and to predict the risk of complications.There are a large number of tools for diagnosing frailty, but not all of them can be used or validated in the ICU (intensive care unit). The need for a tool that is robust, reliable, reproducible and quick to use means that the CFS (Clinical Frailty Scale) a good tool for screening for frailty, particularly in intensive care. It predicts mortality in intensive care and in hospital, regardless of age. However, it requires the cooperation of the patient or the patient's family, and relies on a subjective approach to the patient's state of health by the clinician. This is why, in recent years, new objective tools for diagnosing frailty have been developed, based in particular on anthropometric measurements. The scanographic cross-sectional area of the psoas muscle appears to correlate well with fragility scales in the literature and is an independent risk factor for mortality.

Ultrasound depth of the quadriceps muscle is an easy, rapid and objective measure of the patient's muscle reserves. In the preoperative situation, this measurement correlates with fragility scales and is a risk factor for postoperative morbidity.

We propose to evaluate the diagnostic performance of bilateral ultrasound depth of the quadriceps femoris in comparison with the CFS scale to differentiate frail and non-frail patients in the intensive care unit.

Knowing whether the patient is fragile or not, quickly and objectively, can help the doctor, among other things, to define a reasonable level of therapeutic commitment for the patient and his or her pathology.

to define a reasonable level of therapeutic commitment for the patient and his or her pathology.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 65 or over
* admitted to intensive care or the outpatient department for less than 24 hours
* with an abdominal CT scan less than 30 days prior to admission OR who are scheduled for an scheduled for a routine abdomino-pelvic CT scan within the first 24 hours of admission

Exclusion Criteria:

* Neuromuscular disease
* Lower limb amputation
* Paraplegia > 24 hours before admission
* Clearly infected, burnt or lacerated ultrasound site.
* Guardianship or curatorship
* Opposition of the patient or his/her trusted support person or relative
* Abdominal and pelvic CT scan not available in the previous month and not scheduled within the first 24 hours of treatment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Any patient aged 65 or over admitted to intensive care or the emergency department who meets the eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Bilateral ultrasound depth of the quadriceps femoris muscle | 24 hours
  Bilateral ultrasound depth of the quadriceps femoris muscle: The ultrasound consists of 3 measurements per side of the thickness of the rectus femoris muscle. The ultrasound loops will be recorded on an ultrasound machine (GE) after anonymisation.
  The images will be analysed a posteriori by the principal investigator and the associate investigators, experts in ultrasound analysis of this muscle.

IPD SHARING:
Plan to Share IPD: No